CLINICAL TRIAL: NCT02668679
Title: The Effect of Dream Doctors in Children Undergoing Digestive Endoscopic Procedures: Physiological and Biological Assessment of Emotional and Cognitive Consequences
Brief Title: The Effect of Dream Doctors in Children Undergoing Digestive Endoscopic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Sarit Peleg, Head of Pediatric Gastroenterology Unit, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0068-15-EMC
Record Dates: First submitted 2016-01-10; First posted 2016-01-29 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Gastrointestinal Diseases
Keywords: Dream Doctors; Medical Clown; Pediatrics; Sedation; Endoscopy
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Galvanic Skin Response

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Children and their parents with the presence of Dream Doctors (Active Comparator): The DD will use various methods for entertaining the child and alleviate stress . The parents and the children will be given anxiety and satisfaction questionnaires. The children and parents will perform Pre-Pulse inhibition (PPI) test and GSR. In addition, stress hormones will be assessed (cortisol, epinephrine, and norepinephrine) and the following physical indices will be measured: blood pressure, pulse, saturation and body temperature. The amount of drugs given for deep sedation will be evaluated.
  Interventions: Procedure: Sedation of children during gastroscopy with and without the presence of dream doctor; Device: evaluation of stress with PPI and GSR; Biological: blood specimens for stress hormones; Other: Physiological indices for evaluation of stress
- Children and their parents without the presence of DD (Placebo Comparator): No DD during the gastroscopy. The parents and the children will be given anxiety and satisfaction questionnaires. The children and parents will perform Pre-Pulse inhibition (PPI) test and GSR. In addition, stress hormones will be assessed (cortisol, epinephrine, and norepinephrine) and the following physical indices will be measured: blood pressure, pulse, saturation and body temperature. The amount of drugs given for deep sedation will be evaluated.
  Interventions: Procedure: Sedation of children during gastroscopy with and without the presence of dream doctor; Device: evaluation of stress with PPI and GSR; Biological: blood specimens for stress hormones; Other: Physiological indices for evaluation of stress

INTERVENTIONS:
Procedure: Sedation of children during gastroscopy with and without the presence of dream doctor — children and their parents with and without the presence of DD upon arrival to the Gastroenterology institute and throughout the induction of sedation, gastroscopy and recovery.
  Other Names: dream doctor
Device: evaluation of stress with PPI and GSR — evaluation of stress in children undergoing gastroscopy with sedation with and without the presence of a dream doctor by measurement of PPI and GSR
  Other Names: PPI GSR
Biological: blood specimens for stress hormones — evaluation of stress in children undergoing gastroscopy with sedation with and without the presence of a dream doctor by measurement of stress hormones.
  Other Names: stress hormones
Other: Physiological indices for evaluation of stress — evaluation of stress in children undergoing gastroscopy with sedation with and without the presence of a dream doctor by measurement of blood pressure, pulse, saturation and body temperature.
  Other Names: physiological indices

SUMMARY:
Background: Performance of endoscopy in children requires more patience, experience, and expertise than in adults. The anxiety of the children is related to parent's separation, loss of self-control, unknown surroundings and strange people that are taking care of them, and frequently unpleasant or even painful procedures. Painful and frightening procedures in children have been shown to result in short-term physiologic changes and long-term behavioral changes. The response to unpleasant stimuli with stress and fear may be exaggerated in children and experienced as pain. Most infants and children and many teenagers need deep sedation or light general anesthesia to complete a successful and safe procedure. Induction of general anesthesia is a stressful procedure itself. Strategies to reduce preanesthesia anxiety include pharmacologic and non-pharmacologic interventions.

However, this evidence is based mainly on self reports rather than objective measurements. Therefore, objective and non-invasive measurements to be utilized in the current study, should provide an assessment tools regardless the children's age.

Multiple studies, beginning in the 1970's, have shown that humor has many positive effects on physical and mental health and well-being. Previous investigations have reported that humor has beneficial effects on the immune system, stress related to potentially fatal illnesses, pain tolerance, and mental functions.

Dream doctors (DDs) are professional medical clowns or stage artists, who received training specifically to understand medical patient's need and to give the patient adjuvant therapy during hospital admissions or ambulatory treatment.The Israel dream doctors project, integrates professional medical clowning into the medical services provided at Israeli hospitals.Studies already proved that presence of medical clowns significantly reduces the level of anxiety during induction of anesthesia in children. Hypothesis of the study: 1) DDs lessen the level of anxiety and attention impairment in children undergoing gastroscopies. 2) DDs improve the satisfaction of children and their parents during gastroscopies.

The aim of this study is: 1) To explore the influence of DDs on the satisfaction of children and their parents undergoing gastroscopy, utilizing questioners. 2) To explore the effects of DDs on anxiety and attention of children and their parents, undergoing gastroscopies by means of GSR, startle response and pre-pulse inhibition (PPI) tests, as well as , and measuring anxiety-related biologic indices.

DETAILED DESCRIPTION:
The effect of Dream Doctors in children undergoing digestive endoscopic procedures: Physiological and biological assessment of emotional and cognitive consequences.

Background: Since the advent of pediatric gastrointestinal endoscopy in the early 1970's, there has been a remarkable increase in the number of diagnostic and therapeutic procedures performed in infants and children. Performance of endoscopy in children requires more patience, experience, and expertise than in adults. The anxiety of the children is related to parent's separation, loss of self-control, unknown surroundings and strange people that are taking care of them, and frequently unpleasant or even painful procedures. Painful and frightening procedures in children have been shown to result in short-term physiologic changes and long-term behavioral changes. The response to unpleasant stimuli with stress and fear may be exaggerated in children and experienced as pain. Most infants and children and many teenagers need deep sedation or light general anesthesia to complete a successful and safe procedure. Induction of general anesthesia is a stressful procedure itself. Strategies to reduce preanesthesia anxiety include pharmacologic and non-pharmacologic interventions.

However, this evidence is based mainly on self reports rather than objective measurements. Therefore, objective and non-invasive measurements to be utilized in the current study, should provide an assessment tools regardless the children's age.

Multiple studies, beginning in the 1970's, have shown that humor has many positive effects on physical and mental health and well-being. Previous investigations have reported that humor has beneficial effects on the immune system, stress related to potentially fatal illnesses, pain tolerance, and mental functions.

Dream doctors are professional medical clowns or stage artists, who received training specifically to understand medical patient's need and to give the patient adjuvant therapy during hospital admissions or ambulatory treatment. Laughter has physiological effects on different body mechanisms and it affects the cardiovascular system (decreasing heart rate and blood pressure), strengthens the immune system, and lowers level of stress hormones like Norepinephrine. Humor can also help in strengthening the bond between therapist and patient and reduce stress and anxiety and enhance recovery. The Israel dream doctors project, integrates professional medical clowning into the medical services provided at Israeli hospitals. The DDs are part of the multidisciplinary staff, principally but not only, in pediatric wards. Studies already proved that presence of medical clowns significantly reduces the level of anxiety during induction of anesthesia in children. In the pediatric ward in Afula Medical Center, the investigators have experience with DDs for preparing children to kidney scans.

Pre-Puls Inhibition PPI A computerized human startle response monitoring system (SR-HLAB STARTLE REFLEX, San Diego Instruments, San Diego, CA) was used to deliver acoustic startle stimuli via headphones and record and score the corresponding electro myographic activity from the orbicularis oculi muscle. Two disposable electrodes (sensor area 12 mm2) were placed approximately 0.75-1cm below the pupil on the orbicularis oculi muscle and 3rd reference electrode on the mastoid bone. The skin area at the electrode site was cleaned with a cotton swab saturated with rubbing alcohol, then prepared by gently rubbing a small amount of EEG & ECG Skin Prepping Gel (Signa Gel- Parker Laboratories Inc., Fairfield, New jersey, USA), and cleaned again with a cotton swab.

The session (a total of 56 trials) is started with 3 min acclimatization period with a 60 dB background noise level that is delivered continuously throughout the test session. The session is comprised from two blocks. block1: comprised from randomly delivered six trials of single 40 msec 120 dB "pulse alone" startle stimuli in order to evaluate the startle response, ten "pre" stimuli (at 74, 78, 82, 86 or 92 dB), and thirty "pre pulse" trials that consisted of a single 120 dB pulse preceded (120 msec inter-stimulus-interval) by a 20 msec pre pulse of 14, 18, 22, 26 or 32 dB above background (i.e., 74, 78, 82, 86 or 92 dB). Block1 trials were delivered on average 20 sec inter-trial-interval ITI (15-25 sec, total 46 trials). Block2: comprised of the last ten trials of "pulse alone" startle, at fixed 2 sec ITI in order to evaluate a measure of habituation in response to repeated delivery of the startling stimuli. Finally, prepulse inhibition (PPI) was calculated as the percent of the habituated response as follows [100-(max response to "pre pulse" trial / max response to "pulse alone" trial X 100)]

GSR - Galvanic Skin Response Electrodermal activity will be measured by the differences of the skin conductivity. Two 5 mm electrodes will be placed on fingers 2 and 4 of the non-dominant hand. The electrodes will be connected to sensor and amplifying receiver with a 10Hz sampling rate.

Different portions of the skin can show differences in conductivity, due to sweat related to stress. Thus, measuring the skin conductivity of the non-dominant hand was shown to reduce this variability.

Hypothesis of the study: 1) DDs lessen the level of anxiety and attention impairment in children undergoing gastroscopies. 2) DDs improve the satisfaction of children and their parents during gastroscopies.

The aim of this study is: 1) To explore the influence of DDs on the satisfaction of children and their parents undergoing gastroscopy, utilizing questioners. 2) To explore the effects of DDs on anxiety and attention of children and their parents, undergoing gastroscopies by means of GSR, startle response and pre-pulse inhibition (PPI) tests and measuring anxiety-related biologic indices.

Patients and Methods: This randomized, controlled study will be conducted with children undergoing deep sedation during pediatric upper gastrointestinal endoscopies in the Gastroenterology institute of the Emek Medical Center,Afula, Israel. One hundred children (age 1-18 years) scheduled to undergo deep sedation and elective gastroscopy will be enrolled. During enrollment, the potential clown involvement will be explained to parents. Patients will be assigned to one of two groups: Group 1:children and their parents with the presence of DD upon arrival to the Gastroenterology institute and throughout the induction of sedation, gastroscopy and recovery. Group 2: children and their parents undergoing gastroscopy with deep sedation without the presence of a DD.

The randomization process: In Afula Medical Center, the investigators perform gastroscopies weekly. During the study period the investigators will perform the gastroscopies one week with the DD and one week without the DD.The patients will not be aware to that fact that in some weeks the DD is participating during the sedation induction in some of the patients (every other week). The DD will use various methods for entertaining the child and alleviate stress according to the child's age. The parents and the children will be given anxiety questioners to fill before the induction of sedation. At the end of the gastroscopy the parents and the children will be given satisfaction questioners. The children will perform Pre-Pulse inhibition (PPI) test and GSR before and after the gastroscopy to assess physiological and biological emotional and cognitive consequences. The parents will perform PPI test and GSR before, during and after the gastroscopy (no caffeine or nicotine consumption will be allowed 30min before examination). The anesthesiologist and the nurse at the recovery room will fill a questioner evaluating the behavior of the child during the induction of sedation and awakening. While inserting an IV line blood spots will be taken for stress hormones: cortisol, epinephrine, and norepinephrine. The following physical indices will be measured: blood pressure, pulse, saturation and body temperature. The amount of drugs given for deep sedation will be evaluated.

The current study hold two major innovativeness: (a) The effects of DD as part of the medical team in gastroscopy in children. (b) The physiological and biological evaluation of the emotional and cognitive consequences in children and their parents during gastroscopy.

Statistical analysis:

The study design is Mixed design (2X3), with DD as between subject factor (with or without DD) and stage of treatment as within subject factor (prior, during and after gastroscopy examination).Thus, we will conduct a Two-Way ANOVA (2X3) with post hoc Tukey's test. Significant interactions will be further analyzed with One-Way ANOVA. Moreover to relate physiological and biological measurement to questioner items, Pearson's correlations will be calculated.

The study schedule:

1. Recruitment: 1.5 year
2. Study period: for each patient the study will be held during the day of gastroscopy.
3. Examination of blood serum by ELISA: 3 months.

3. Analysis of results: three months 4. Targeted date as to completion of project: two years from the study beginning.

Project staff:

1. Dr Peleg Sarit - Board certified in Pediatrics and Pediatric Gastroenterology and Nutrition.
2. Dr Rinawi Firas - Board certified in Pediatrics and Pediatric Gastroenterology and Nutrition.
3. Dr Efrat Rachel - Board certified in Anesthesiology and Pediatrics.
4. Professor Avital Avi - Behavioral Neuroscience Lab, Head.
5. Mrs Lazimi Ilanit - Pediatric and Pediatric Gastroenterology nurse.
6. Mr Yaron (Sancho) Goshen - Experienced DD.
7. Mrs Yaara Tirosh Kamienchick - Research coordinator. Institutional overview: Dr Peleg Sarit, Pediatric Gastroenterology Unit, Emek Medical Center, Shderot Itzhak Rabin 21 Afula, 18101, Israel Phone: +972-4-6494104 Fax: +972-4-6495532 Email: Peleg_sa@clalit.org.il

Ethics:

The study will be conducted according to the ethical principles of the Declaration of Helsinki. Informed consent will be obtained following explicit description of the study outline and alternatives for participation. It will be made clear that declining to participate in the study will not jeopardize, in any way, the quality of care received. The signed consent will be filed in the patient's medical record. The principal investigators will have full access to the data prior to publication. CRFs will be identified and coded by study number and initials only.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years undergoing gastroscopy.
* Informed consent of the parents

Exclusion Criteria:

* Developmental delay or neurologic disease
* Children who underwent endoscopy in the past
* Parents that don't agree to participate in the study
* ASA≥3
* Children or parents hearing problem.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Level of anxiety in children undergoing gastroscopies measured by biological indices (blood pressure) | Up to 12 hours during the day of gastroscopy for each patient.
  The following physical indices will be measured: blood pressure (mmHG)
Level of anxiety in children undergoing gastroscopies measured by biological indices (pulse) | Up to 12 hours during the day of gastroscopy for each patient.
  The following physical indices will be measured: pulse per minute
Level of anxiety in children undergoing gastroscopies measured by biological indices (saturation) | Up to 12 hours during the day of gastroscopy for each patient.
  The following physical indices will be measured: saturation meaning level of oxygen in blood with pulse oximeter in units
Level of anxiety in children undergoing gastroscopies measured by biological indices (body temperature) | Up to 12 hours during the day of gastroscopy for each patient.
  The following physical indices will be measured: body temperature in celsius degrees
Level of anxiety in children undergoing gastroscopies measured by biological indices (sedation drug level) | Up to 12 hours during the day of gastroscopy for each patient.
  The following physical indices will be measured:The amount of drugs given for deep sedation will be evaluated, in milligrams per kilogram body weight.
level of anxiety in children undergoing gastroscopies and their parents measured by PPI | Up to 12 hours during the day of gastroscopy for each patient.
  The investigators would use a monitoring device that would assess startle reflex reaction measured by blinking of the eye. Monitoring would be done with electrodes of EMG device that would be located on orbicularis oculi muscle and will monitor response. Startle reflex response (anxiety)- Assessed by millivolts registered by electromyography (EMG) electrodes.
level of anxiety in children undergoing gastroscopies and their parents measured by GSR | Up to 12 hours during the day of gastroscopy for each patient.
  The investigators would use a monitoring device that would assess physiological reactivity by measurement of skin conductance (galvanic skin response).

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Peleg, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel

REFERENCES:
- [Result] Tolia V, Peters JM, Gilger MA. Sedation for pediatric endoscopic procedures. J Pediatr Gastroenterol Nutr. 2000 May;30(5):477-85. doi: 10.1097/00005176-200005000-00003. No abstract available. PMID 10817274
- [Result] Soker Z. Play and Learning: What really children wan't to learn through play? 'Megamot' (Trends) for research. Behav. Sci.1993; 34:497-520.
- [Result] Puder C. The healthful effects of laughter. CYC-Net 2003; 55:32-42.
- [Result] Golan G, Tighe P, Dobija N, Perel A, Keidan I. Clowns for the prevention of preoperative anxiety in children: a randomized controlled trial. Paediatr Anaesth. 2009 Mar;19(3):262-6. doi: 10.1111/j.1460-9592.2008.02903.x. Epub 2008 Dec 23. PMID 19143948
- [Result] Vagnoli L, Caprilli S, Messeri A. Parental presence, clowns or sedative premedication to treat preoperative anxiety in children: what could be the most promising option? Paediatr Anaesth. 2010 Oct;20(10):937-43. doi: 10.1111/j.1460-9592.2010.03403.x. PMID 20849499